CLINICAL TRIAL: NCT01659489
Title: Blood and Serum Markers in Patients Operated for Suspected Ovarian Torsion
Brief Title: ADnexal TOrsion Markers Study
Acronym: ATOMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Roy Mashiach, M.D., Senior Physician, Sheba Medical Center
Other Study IDs: SHEBA-12-9605-RM-CTIL
Record Dates: First submitted 2012-07-31; First posted 2012-08-07 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Adnexal Torsion; Laparoscopy
Keywords: adnexal torsion; laparoscopy
MeSH Terms: conditions — Ovarian Torsion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum will be frozen for evaluation
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- women undergoing laproscopy fo rsuspected adnexal torsion

SUMMARY:
Adnexal torsion , is a severe, though uncommon gynecological emergency, with a prevalence of 2.7-3%. The need for prompt diagnosis and treatment in order to save ovarian tissue has been realized a long time ago. A marker that will aid in the diagnosis of torsion and prevent missed diagnosis and unecessary loss of ovarian tissue, while not increasing the rate of unecessary laparoscopic interventions is much needed. To our knowledge, such marker has not been found. The purpose of this study is to find a marker using blood/serum from patients undergoing laparoscopy for suspected ovarian torsion

DETAILED DESCRIPTION:
Adnexal torsion, is a severe, though uncommon gynecological emergency, with a prevalence of 2.7-3% (Taskin 1998; Hibbard1985;Burnett 1988). Torsion commonly occurs in children and women of childbearing age (Haskins 1986).

The need for prompt diagnosis and treatment in order to save ovarian tissue has been realized a long time ago (Ben-Arie 1995). The accuracy of clinical diagnosis is low, with a false negative rate of up to 56% (Cohen 2001, Bar-On 2010,Mashiach 2010). Doppler ultrasound tests, do not "necessarily exclude an ovarian torsion; in fact, "the diagnosis of" torsion is missed in 60% of cases, and time to diagnosis in these cases is delayed" (Pena 2001).

Therefore there is a need for a marker that will aid in the diagnosis of torsion and prevent missed diagnosis and unecessary loss of ovarian tissue, while not increasing the rate of unecessary laparoscopic interventions, which are often performed in an emergency setup, by unqualified personnel.

To our knowledge, such marker has not been found. The purpose of this study is to find a marker, or marker combination, using blood/serum from patients undergoing laparoscopy for suspected ovarian torsion study type: a prospective, controlled, blind study study population: 200 women undergoing laparoscopy for ovarian torsion

ELIGIBILITY:
Inclusion Criteria:

* women undergoing laparoscopy for suspected ovarian torsion

Exclusion Criteria:

* elevated liver enzymes
* suspected ovarian malignancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 200 women undergoing laparoscopy for suspected ovarian torsion in a tertiary referral center
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-08; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Serum level of blood proteins (complete list available by direct contact)will be measured before and after ovarian detorsion, and will be compared to those taken from patients who were underwent diagnostic laparoscopy for suspected ovarian torsion. | Blood will be withrawed before and within 12 hourse after the surgery. The results will be analysed after recruitment and blood withrawal is finished. not later than three years after the begining of the trial

CONTACTS AND LOCATIONS:
Locations (1):
- The chaim sheba medical center,Tel Hashomer, Ramat Gan, Israel